CLINICAL TRIAL: NCT03188744
Title: Impact of Cancer Treatment on the Pelvic Floor Function in Survivors of Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Aline Moreira Ribeiro, MSc., University of Sao Paulo
Other Study IDs: 5557/2017
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Cervical Cancer; Pelvic Floor Disorders; Surgery; Radiotherapy; Complications; Chemotherapy Effect
Keywords: Cervical cancer; Pelvic floor muscles; Physiotherapy; Quality of life
MeSH Terms: conditions — Uterine Cervical Neoplasms; Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Patients with CC with PFMD.
  Interventions: Other: Assessment of the pelvic floor function; Other: Questionnaire application
- Group 2: Patients with CC without PFMD.
  Interventions: Other: Assessment of the pelvic floor function; Other: Questionnaire application
- Group 3: Patients without CC with PFMD.
  Interventions: Other: Assessment of the pelvic floor function; Other: Questionnaire application
- Group 4: Patients without CC without PFMD.
  Interventions: Other: Assessment of the pelvic floor function; Other: Questionnaire application

INTERVENTIONS:
Other: Assessment of the pelvic floor function — Vaginal palpation and perineometry.
Other: Questionnaire application — Questionnaires: EORTC, WHOQoL-BREF, PFID-20; PSIQ-12 and PFIQ-7.

SUMMARY:
Introduction: Pelvic floor muscle dysfunctions (PFMD) represent an important public health problem that manifests itself through lower urinary tract symptoms (LUTS), anorectal and sexual dysfunction. PFMD is a common problem in cervical cancer survivors (CC) with a negative impact on quality of life (QoL). Objective: This study aims to evaluate the effect of oncological treatment on the function of pelvic floor muscles (PFM) of survivors of CC. Methods: Patients diagnosed with CC, of any stage, histology and degree, accompanied by the Oncology Gynecology Service of the Hospital das Clínicas of the Medical School of Ribeirão Preto at the University of São Paulo, will be studied in the period between 2004 and 2014. Four study groups will be formed: (1) Patients with CC with PFMD; (2) Patients with CC without PFMD; : (3) Patients without CC with PFMD; (2) Patients without CC without PFMD. Non-cancer patients will be recruited into the community. For the analysis of the prevalence of PFMD will be applied to the discomfort Questionnaire on pelvic floor (IDPE-20) for evaluation of pelvic organ prolapse (POP) complaints, anorectal symptoms and urinary incontinence, and the Sexual Questionnaire for urinary incontinence and pelvic organ prolapse (PISQ -12) for evaluation of sexual function. Both questionnaires have already been validated for the Portuguese language and are specific for women with PFMD. The pelvic floor impact questionnaire (PFIQ-7) will also be applied to assess the impact of PFMD on quality of life, daily living activities and emotional health. For the evaluation of general QOL, the EORTC questionnaire QLQ-C30 and its specific module for patients with CC, QLQ-CX24 will be used. The evaluation of PFM function will include vaginal palpation (Modified Oxford Scale) and perineometry (Peritron).

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with CC; No distinction as to age, race, scholarity and religion; Women in follow-up at Clinical Hospital of Medical School of Ribeirão Preto of University São Paulo.

Exclusion Criteria:

* Women who did not complete the proposed cancer treatment; Women who presented CC as the second malignant neoplasm; Pregnant women; Failure to respond to the proposed questionnaires.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with CC with and without PFMD and women without CC with and without PFMD.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-01-02 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor muscles function | Four months
  Evaluated through vaginal palpation and perineometry.

SECONDARY OUTCOMES:
Quality of life in the pelvic floor muscles dysfunction. | Four months
  Evaluated through application of the questionnaire PFIQ-7.
Prevalence of the pelvic floor muscles dysfunction. | Four months
  Evaluated through application of the questionnaires PSIQ-12 and PFID-20.
Overall quality of life. | Four months
  Evaluated through application of the questionnaires EORTC QLQ-C30 and its specific module for patients with CC, QLQ-CX24 and the WHOQoL-BREF questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Harley Oliveira, PhD, Study Director — University of Sao Paulo
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greimel ER, Kuljanic Vlasic K, Waldenstrom AC, Duric VM, Jensen PT, Singer S, Chie W, Nordin A, Bjelic Radisic V, Wydra D; European Organization for Research and Treatment of Cancer Quality-of-Life Group. The European Organization for Research and Treatment of Cancer (EORTC) Quality-of-Life questionnaire cervical cancer module: EORTC QLQ-CX24. Cancer. 2006 Oct 15;107(8):1812-22. doi: 10.1002/cncr.22217. PMID 16977652
- [Result] Arouca MA, Duarte TB, Lott DA, Magnani PS, Nogueira AA, Rosa-E-Silva JC, Brito LG. Validation and cultural translation for Brazilian Portuguese version of the Pelvic Floor Impact Questionnaire (PFIQ-7) and Pelvic Floor Distress Inventory (PFDI-20). Int Urogynecol J. 2016 Jul;27(7):1097-106. doi: 10.1007/s00192-015-2938-8. Epub 2016 Jan 19. PMID 26782099
- [Result] Santana GW, Aoki T, Auge AP. The Portuguese validation of the short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12). Int Urogynecol J. 2012 Jan;23(1):117-21. doi: 10.1007/s00192-011-1505-1. Epub 2011 Jul 28. PMID 21796471
- [Result] Hazewinkel MH, Sprangers MA, Taminiau-Bloem EF, van der Velden J, Burger MP, Roovers JP. Reasons for not seeking medical help for severe pelvic floor symptoms: a qualitative study in survivors of gynaecological cancer. BJOG. 2010 Jan;117(1):39-46. doi: 10.1111/j.1471-0528.2009.02411.x. PMID 19874292